CLINICAL TRIAL: NCT06040398
Title: The JUMPSTART Program: Encouraging Early Mobilization and Optimizing Recovery of TAVR Patients' Post-hospital Discharge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Edwards Lifesciences (Industry); McMaster University (Other)
Responsible Party: Principal Investigator, Madhu K. Natarajan, Interventional and Structural Cardiologist; Professor, McMaster University, Hamilton Health Sciences Corporation
Organization: McMaster University (Other)
Other Study IDs: 15474
Record Dates: First submitted 2023-07-12; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement
Keywords: early mobilization; exercise program; cardiac care
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TAVR Patients: All outpatients undergoing TAVR and managed through the overnight-model pathway at the Hamilton General Hospital will be eligible for participation.
  Interventions: Behavioral: JUMPSTART exercise program

INTERVENTIONS:
Behavioral: JUMPSTART exercise program — The intervention is an early mobilization protocol (JUMPSTART). Four interactive exercise videos, at different intensity levels, include a variety of stretches and exercises designed to improve the full body mobilization of post-TAVR patients. Videos have been developed in consultation with a physiotherapist and cardiac rehabilitation specialist and have been piloted for initial acceptability by patients at the Hamilton General Hospital. The videos will be freely accessible to all eligible patients and their caregivers (regardless of participation in the research study) online (www.hhscebi.ca/projects/jumpstart). A written version of the exercise program, with photographs and detailed instructions, will also be made available. Additional exercise videos will be developed based on patients' needs and feedback received.

SUMMARY:
A virtual, self-directed, and tailored early mobilization program called JUMPSTART, that aims to bridge cardiac rehabilitation intake for post-TAVR patients has been developed at the Hamilton General Hospital. The program includes a series of exercise videos at varying levels of intensity, designed for patients to follow at home, post-discharge. JUMPSTART is currently being offered as part of clinical care. In this new pilot study, the study team plans to develop and test new strategies to optimize recruitment and participation, develop additional JUMPSTART materials and evaluate outcomes through follow-up surveys and registry/administrative data at Hamilton General Hospital.

DETAILED DESCRIPTION:
Post-TAVR patients who have successfully completed a pre-discharge ambulation assessment and are deemed eligible for discharge will be eligible to participate. Potential participants will be introduced to the study in the pre-TAVR clinic by the nurse practitioner or their delegate. Participants who agree to be contacted for research purposes will provide written consent in the pre-TAVR clinic when they meet with the nurse practitioner. Confirmation of eligibility for the research study will be conducted post-TAVR by the nurse practitioner. The JUMPSTART program will be offered to all eligible patients as part of standard clinical care, regardless of their consent to participate in the research study. No data will be collected for the purposes of the research study from patients who do not provide consent. The primary outcomes will be adoption (the number of eligible post-TAVR patients who participate in the JUMPSTART early mobilization program), and a preliminary comparison of quality of life (measured using the Toronto Aortic Stenosis Quality of Life Questionnaire) between people who do and do not participate in the JUMPSTART program.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients who have undergone a TAVR procedure at the Hamilton General Hospital
* Patients who are managed through the overnight-model pathway
* Patients who successfully completed ambulation assessment
* Patients who are deemed eligible for discharge

Exclusion Criteria:

* Patients who are hospitalized after the procedure (inpatients)
* Patients who had an axillary approach for TAVR
* Patients who had a pacemaker temporarily left in at the end of case, and
* Patients who received a permanent pacemaker in the last month

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population of post-TAVR patients is growing larger and ranges in age from 65 to 95 years.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness (quality of life) | Baseline and 3 months post-TAVR procedure.
  Changes in Toronto Aortic Stenosis QoL Questionnaire (TASQ) scores will be compared among study participants who did the JUMPSTART program, and those that didn't. The TASQ consists of 16 statements. Most statements are answered via 7-point Likert scale, where a higher score represents worse outcomes.
Adoption | 14 days post-TAVR procedure.
  Number of eligible patients who participate in the JUMPSTART program.
Adoption | 3 months post-TAVR procedure.
  Number of eligible patients who participate in the JUMPSTART program. Target = 70% adoption rate.

SECONDARY OUTCOMES:
Reach | 12 months (post-study start date).
  Assessed by dividing the total eligible number of TAVR patients who agree to enter the JUMPSTART program by the total eligible number of TAVR patients who underwent the TAVR procedure at the Hamilton General Hospital.
Effectiveness (cardiac rehab attendance) | 3 months post-TAVR procedure.
  Measurement of the percentage of post-TAVR patients who have attended a cardiac rehab orientation session by 3 months post-TAVR procedure.
Effectiveness (acceptability) | 14 days and 3 months post-TAVR procedure.
  Acceptability will be measured by self-reported questionnaire in consenting participants, administered via telephone interview or online survey (REDCap). Participants are asked to provide their level of satisfaction with the exercise videos and instructional handout on a scale of 1-7, where 1 = very unsatisfied and 7 = very satisfied.
Effectiveness (feasibility) | 14 days and 3 months post-TAVR procedure.
  Feasibility will be measured by self-reported questionnaire in consenting participants, administered via telephone interview or online survey (REDCap). Participants are asked about ease in following the exercise videos, and challenges associated with doing the exercises.
Adoption (barriers and facilitators) | 14 days and 3 months post-TAVR procedure.
  Barriers and facilitators will be assessed by questionnaire administered via telephone interview or online survey (REDCap). No response scales are used, the data collected is qualitative in nature. Implementation strategies will be tailored to these barriers and facilitators using an iterative process.
Implementation (fidelity) | Assessed at 4 months (post-study start date), 8 months, and 12 months.
  Meetings/focus groups with research team and hospital staff to review whether implementation has taken place as planned (e.g., fidelity of the recruitment process, data collection), and to discuss pre-discharge testing and whether patients are given JUMPSTART materials both at the pre-TAVR clinic and prior to discharge.
Maintenance | Assessed at 4 months (post-study start date), 8 months, and 12 months.
  Meetings/focus groups with research team to review study participation rates and to discuss barriers to participation. Program sustainability and plans for imbedding the program into routine care/practice will also be discussed.

CONTACTS AND LOCATIONS:
Overall Officials: Madhu K Natarajan, MD, Principal Investigator — Hamilton Health Sciences and McMaster University
Locations (1):
- Hamilton Health Sciences (McMaster Children's Hospital and Hamilton General Hospital), Hamilton, Ontario, Canada